CLINICAL TRIAL: NCT05553119
Title: Home-based Pulmonary Rehabilitation and Health Coaching in Bronchiectasis
Brief Title: A Study of Home-based Pulmonary Rehabilitation and Health Coaching to Treat Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Other Study IDs: 22-004626; 5K24HL138150-05 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home-based Pulmonary Rehabilitation and Health Coaching: Subjects with symptomatic bronchiectasis (CAT score ≥10) will receive a 12-week intervention with home-based pulmonary rehab (PR).
  Interventions: Behavioral: Home Rehabilitation Monitoring System; Behavioral: Health coaching calls

INTERVENTIONS:
Behavioral: Home Rehabilitation Monitoring System — Established home-based pulmonary rehab system consists of three commercial devices (Garmin Vívofit™ activity monitor, Nonin 3150 WristOx2® Pulse Oximeter, Android tablet) and two software applications for telemonitored home pulmonary rehabilitation.
Behavioral: Health coaching calls — Coaching calls based on motivational interviewing principles will occur weekly for twelve weeks following a standard protocol, lasting no more than 5-10 minutes.

SUMMARY:
The purpose of this study is to gather information on the effectiveness on a home-based pulmonary rehabilitation in patients with bronchiectasis.

DETAILED DESCRIPTION:
The purpose of this study is to gather information on the effectiveness on a home-based pulmonary rehabilitation in patients with bronchiectasis. We hope that by participating in home-rehab that patients with bronchiectasis will become more physically active in their daily lives.

Pulmonary Rehabilitation in a medical center has proven to have a positive impact on physical activity and shortness of breath in patients with chronic lung disease. However, travel and access can make going to a center difficult.

Study participation involves completing gentle flexibility exercises and walking practice using a provided computer tablet, pulse oximeter and an activity tracker for 12 weeks. During that time, you will talk to a health coach once a week on the phone. At the end of the 12 weeks, someone will call you and ask you questions about your experience with the home-based rehab. Health Coaching calls will be recorded so that it can later be transcribed. All identifying information will be removed and the answers will be lumped together.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of non-cystic fibrosis bronchiectasis (primary inclusion criteria) ,confirmed by records, that are symptomatic.
* Ability to communicate in English.

Exclusion Criteria:

* Inability to walk (orthopedic/neurologic/cardiac limitation causing immobility).
* Cognitive impairment or inability to understand and follow instructions.
* Traditional PR completed within 3 months of study recruitment.
* Hospice or end-of-life care at the time of screening.
* Acute exacerbation at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a medical diagnosis of bronchiectasis being see in the Mayo Clinic Bronchiectasis Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported quality of life | Baseline, after completion of the 12-week intervention.
  As defined by the COPD Assessment Test (CAT). The CAT is a validated tool for measuring health status in patients with bronchiectasis and is divided into eight domains of cough, mucous production, chest tightness, shortness of breath with activity, activity limitation at home, confidence leaving home, sleep quality, and energy. A lower score suggests no health-related quality of life (HRQL) impairment, while the maximum score of 40 represents significant impact.

SECONDARY OUTCOMES:
Physical activity | 12 weeks
  As measured by number of steps per 24-hr period.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials